CLINICAL TRIAL: NCT00656708
Title: Kerlix AMD Gauze Study In A Burn Trauma Unit and Its Effect on Healthcare Associated Infections in Burn Patients
Brief Title: Kerlix Gauze Study in a Burn Trauma Unit and Its Effect on Healthcare Associated Infections in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucy A Wibbenmeyer (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor-Investigator, Lucy A Wibbenmeyer, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 200703800
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2009-08

CONDITIONS: Burns; Wounds
Keywords: Burns; Wounds; Healthcare associated infections; MRSA; VRE
MeSH Terms: conditions — Burns; Wounds and Injuries; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- PB (Experimental): All patients admitted to the burn unit during the prospective portion (interventional portion) of the study who have open wounds will have Kerlix AMD applied to their wounds; only those patients consenting to the study will have data abstracted.
  Interventions: Other: Kerlix AMD gauze

INTERVENTIONS:
Other: Kerlix AMD gauze — Use Kerlix AMD gauze as the wound dressing for the entire burn unit
  Other Names: Kerlix Gauze

SUMMARY:
The purpose of this study is to determine whether Kerlix AMD gauze will decrease the incidence of healthcare associated infections in burn patients. Kerlix AMD gauze will be applied to all patients with open wounds admitted to the burn unit during the prospective portion of the study. All consenting patients will be assessed for hospital associated infections and outcomes. We hypothesis that burn patients will have a decreased number of hospital associated infections compared to historical controls.

DETAILED DESCRIPTION:
Infection continues to cause significant morbidity in burn patients. Among critically ill patient populations, burn patients have some of the highest rates of device related infections. The loss of integument accompanied with the immunosuppression of the burn injury makes burn patients highly susceptible to infection. Despite the use of daily hydrotherapy, topical antimicrobials and early surgical intervention, sepsis frequently occurs. The burn wound is a major source of nosocomial infections. The standard burn wound dressing at UIHC consists of silver sulfadiazine cream and an outer dressing of woven, porous gauze. A newer version of woven, porous gauze, KERLIX AMD, Covidien, Mansfield, MA, offers additional protection for wounds that require dressing or packing. KERLIX AMD differs from plain gauze only in its impregnation with 0.2% polyhexamethylene biguanide (PHMB). PHMB is chemically related to chlorhexidine gluconate (CHG) which is a biguanide. PHMB has been used as a broad spectrum antiseptic in products such as pool cleaners. Further, PHMB is a broad spectrum biocide that is active against a wide range of pathogens that includes MRSA, VRE, Candida albicans, Pseudomonas aeruginosa, multi-drug resistant Acinetobacter as well as many other pathogens. Clinical exposure is several orders of magnitude less than that associated with acute toxicity (6.46 mg/PHMB/kg v 400 mg PHMB/kg). Clinical use of KERLIX AMD has shown a decrease in wound colonization and a decrease in surgical site infections in multiple wound types. We hypothesize that Kerlix AMD dressing will decrease the incidence of nosocomial infections in our burn patients.

Upon admission to the burn unit, all patients with open wounds will have their wounds dressed with KERLIX AMD Gauze. Patients will then be approached to have their data collected and analyzed for the study. Only patients consenting to the study will have their data collected.

The gauze will be applied directly to all open torso or extremity wounds over a layer of Silver Sulfadiazine immediately after admission to 8JC. The gauze will be used until wounds no longer require dressing. There will be no restriction on the use of topical antibiotics, although Dakin's solution will be restricted. Studies have shown that Dakin's solution deactivates the PHMB.( Tyco Healthcare Group LP) There will be no restriction on the outer layers of the wound dressing or the frequency of dressing changes.

When 108 burn subjects have completed enrollment, the study will be stopped and the data analyzed. Historical infection data will be obtained by reviewing the charts of the last 324 burn patients (with LOS>48 hours) prior to study commencement. Historical data will be compared to the KERLIX AMD gauze study data. All data analyses will be conducted by a biostatistician. Infections will be defined by modified Centers for Disease Control (CDC) criteria.10

ELIGIBILITY:
Inclusion Criteria:

* admitted to the burn unit with a burn or open wound and anticipated to have a length of stay greater than 48 hours

Exclusion Criteria:

* pregnant or nursing women
* wound is considered unsuitable for study dressings as determined by primary physician
* use of Dakin's solution on wound

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the incidence of healthcare associated infections in the study of the acute burn population when using Kerlix AMD gauze as compared to that in matched historical controls when using standard, non-impregnated gauze. | 2 years

SECONDARY OUTCOMES:
Compare the incidence of wound infections between the acute burn study patients and the matched historical control patients. | 2 years
Compare the incidence of healthcare associated infections in the unit when using Kerlix AMD to the previous year using standard gauze. Epidemiology infection rates will be used to compare the incidence of infections. | 2 years
Compare the presence of pathogenic organisms on weekly wound swabs between the acute burn study patients and the matched historical control patients. | 2 years
Compare the nasal MSSA/MRSA colonization between the acute burn study patients and the matched historical control patients. | 2 years
Compare the incidence of rectal VRE colonization between the acute burn study patients and the matched historical control patients. | 2 years
Compare the length of stay per body surface area burned between the acute burn study patients and the matched historical control patients. | 2 years
Compare the antibiotic usage between the acute burn study patients and the matched historical control patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lucy A Wibbenmeyer, MD, Principal Investigator — The University of Iowa Hospitals & Clinics
Locations (1):
- The University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelgren P, Bjornhagen V, Bragderyd K, Jonsson CE, Ransjo U. A prospective study of infections in burn patients. Burns. 2002 Feb;28(1):39-46. doi: 10.1016/s0305-4179(01)00070-5. PMID 11834328
- [Background] Taylor GD, Kibsey P, Kirkland T, Burroughs E, Tredget E. Predominance of staphylococcal organisms in infections occurring in a burns intensive care unit. Burns. 1992 Aug;18(4):332-5. doi: 10.1016/0305-4179(92)90158-q. PMID 1418512
- [Background] Wibbenmeyer L, Danks R, Faucher L, Amelon M, Latenser B, Kealey GP, Herwaldt LA. Prospective analysis of nosocomial infection rates, antibiotic use, and patterns of resistance in a burn population. J Burn Care Res. 2006 Mar-Apr;27(2):152-60. doi: 10.1097/01.BCR.0000203359.32756.F7. PMID 16566558
- [Background] Wurtz R, Karajovic M, Dacumos E, Jovanovic B, Hanumadass M. Nosocomial infections in a burn intensive care unit. Burns. 1995 May;21(3):181-4. doi: 10.1016/0305-4179(95)80005-9. PMID 7794498
- [Background] National Nosocomial Infections Surveillance (NNIS) System Report, Data Summary from January 1992-June 2001, issued August 2001. Am J Infect Control. 2001 Dec;29(6):404-21. doi: 10.1067/mic.2001.119952. No abstract available. PMID 11743489
- [Background] Stone PW, Braccia D, Larson E. Systematic review of economic analyses of health care-associated infections. Am J Infect Control. 2005 Nov;33(9):501-9. doi: 10.1016/j.ajic.2005.04.246. PMID 16260325
- [Background] Mayhall CG. The epidemiology of burn wound infections: then and now. Clin Infect Dis. 2003 Aug 15;37(4):543-50. doi: 10.1086/376993. Epub 2003 Jul 30. PMID 12905139
- [Background] Motta GJ, Milne CT, Corbett LQ. Impact of antimicrobial gauze on bacterial colonies in wounds that require packing. Ostomy Wound Manage. 2004 Aug;50(8):48-62. PMID 15356368
- [Background] Motta GJ, Trigilia D. The effect of an antimicrobial drain sponge dressing on specific bacterial isolates at tracheostomy sites. Ostomy Wound Manage. 2005 Jan;51(1):60-2, 64-6. PMID 15695836
- [Background] Garner JS, Jarvis WR, Emori TG, Horan TC, Hughes JM. CDC definitions for nosocomial infections, 1988. Am J Infect Control. 1988 Jun;16(3):128-40. doi: 10.1016/0196-6553(88)90053-3. PMID 2841893